CLINICAL TRIAL: NCT01973751
Title: Novel Asthma Biomarkers to Predict the Response to Inhaled Corticosteroid
Brief Title: Asthma Biomarkers for Predicting Response to Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Guohua Zhen, MD, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81170022; 30770941
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy controls (No Intervention): Healthy controls who will be studied at baseline and serve as a control group for the bronchoscopy, induced sputum and peripheral blood collection.
- Asthmatics (treatment) (Active Comparator): Steroid-naïve asthma, randomized to inhaled budesonide, 2 puffs (200mcg) twice a day for 8 weeks. These subjects will undergo bronchoscopy and induced sputum collection at baseline, undergo pulmonary function testing and peripheral blood collection at baseline, 4 and 8 weeks after treatment with inhaled corticosteroids.
  Interventions: Drug: Budesonide
- Asthmatics (no treatment) (No Intervention): Steroid-naïve asthmatics randomized to no treatment for 8 weeks. These subjects will undergo bronchoscopy and induced sputum collection at baseline, undergo pulmonary function testing and peripheral blood collection at baseline, 4 and 8 weeks of no treatment.

INTERVENTIONS:
Drug: Budesonide — Inhaled powder of inhaled corticosteroid, 2 puffs (200mcg) twice a day for 8 weeks
  Other Names: Pulmicort
  Arms: Asthmatics (treatment)

SUMMARY:
Novel asthma biomarkers to predict the response to inhaled corticosteroid Brief description: This will be a single center study of asthmatic subjects and healthy controls which will investigate mechanisms underlying different response to inhaled corticosteroid, the mainstay of asthma therapy. Only about half of the asthmatic patients have improved lung function after treatment of inhaled corticosteroid. The investigators hypothesize that there are biomarkers such as epithelial cytokines (IL-25, IL-33, TSLP) in airway tissues or plasma of asthmatic patients which could predict the response of asthmatic patients to inhaled corticosteroid. Finding novel asthma biomarker will help the clinicians to choose the optimal treatment for individual asthmatic patient.

ELIGIBILITY:
Group A:

Inclusion Criteria:

* Male and female subjects between the ages of 18 and 70 years
* No respiratory symptoms
* Normal spirometric value and methacholine PD20 >2.5mg

Group B:

Inclusion Criteria:

* Male and female subjects between the ages of 18 and 70 years
* History of asthma
* No use of oral or inhaled corticosteroids for the treatment of asthma
* No use of leukotriene antagonist for the treatment of asthma
* Hyperreactivity to methacholine (PD20 FEV1 Methacholine < 2.5 mg) and/or ≥12% increase in FEV1 following inhalation of 200μg salbutamol
* Asthma symptoms of episodic cough, wheeze and/or breathlessness

Exclusion Criteria:

* Current or former smokers
* Pregnant women
* Subjects with a history of lung disease other than asthma
* Subjects with a history of a medical disease, which in the opinion of the investigator may put the subject at extra risk from study-related procedures or because the disease may influence the results of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline airway epithelial cytokines expression, FEV1 and methacholine PD20 at 4 and 8 weeks | 8 weeks
  1. The baseline expression of airway epithelial cytokines (IL-25, IL-33, TSLP) and/or Th2 cytokines (IL-4, IL-5, IL-13) in bronchial brushing, bronchial biopsy and peripheral blood in healthy control subjects and asthmatic patients.
  2. Change of forced expiratory volume of the 1st second (FEV1) and accumulated dosage of methacholine provoking a 20% fall of in forced expiratory volume in the first second (FEV1 PD20) of asthmatic patients after treatment with inhaled budesonide or non-intervention for 4 and 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Tongji Hospital, Wuhan, Hubei, China